CLINICAL TRIAL: NCT05002777
Title: A Multicenter, Open-label, Phase IIb Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Rilzabrutinib in Patients With Warm Autoimmune Hemolytic Anemia (LUMINA 2)
Brief Title: Efficacy, Safety and Pharmacokinetics of Rilzabrutinib in Patients With Warm Autoimmune Hemolytic Anemia (wAIHA)
Acronym: LUMINA 2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT17209; U1111-1262-2929 (Registry Identifier: ICTRP); 2023-509441-13 (Registry Identifier: CTIS); 2021-001671-16 (EudraCT Number)
Record Dates: First submitted 2021-08-05; First posted 2021-08-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Warm Autoimmune Hemolytic Anemia (wAIHA)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rilzabrutinib (Experimental): Oral rilzabrutinib 400 mg BID
  Interventions: Drug: rilzabrutinib

INTERVENTIONS:
Drug: rilzabrutinib — Pharmaceutical form: Tablet Route of administration: Oral
  Other Names: PRN1008/SAR444671

SUMMARY:
All participants will receive rilzabrutinib orally. The screening period is up to 28 days, followed by a treatment period of 24 weeks for Part A. Participants who complete Part A and are deemed eligible for Part B can continue in the Core Part B period followed by an Extended Part B period for up to 253 weeks.

There will be a 7-day safety follow-up period after receiving the last dose of study medication either in Part A (for those not eligible for Part B or early terminated) or Part B. In addition, each participant will be asked to attend an EOT-Core Part B visit when the last participant completes 52 weeks in Core Part B. The Extended Part B period will last for up to 253 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a confirmed diagnosis of primary wAIHA or systemic lupus erythematosus (SLE)-associated wAIHA (without other SLE-related manifestations apart from cutaneous and musculoskeletal manifestations)
* Participants who have previously failed to maintain a sustained response after treatment with corticosteroids.
* Eastern Cooperative Oncology Group (ECOG) performance status grade 2 or lower.
* Up-to-date vaccination status as per local guidelines.
* Body mass index (BMI) >17.5 and <40 kg/m2
* All contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Core Part B

* Evidence of treatment efficacy to rilzabrutinib as defined by achieving overall response during Part A.
* Completion of Part A treatment period (24 weeks). Extended Part B
* Completion of Core Part B period.

Exclusion Criteria:

* Clinically significant medical history or ongoing chronic illness that would jeopardize the safety of the participant or compromise the quality of the data derived from his or her participation in the study as determined by the Investigator.
* Participants with medical history of lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for the past 3 years.
* Secondary wAIHA from any cause including drugs, lymphoproliferative disorders (low-count monoclonal B-cell lymphocytosis is allowed), infectious or autoimmune disease, or active hematologic malignancies. Participants with positive antinuclear antibodies but without a definitive diagnosis of an autoimmune disease are allowed.
* Myelodysplastic syndrome.
* Uncontrolled or active HBV infection: Patients with positive HBsAg and/or HBV DNA.
* HIV infection.
* Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days or 5 half-lives, whichever is greater, prior to treatment start.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.

Part B only

* Participants who receive any therapy during Part A known to be active in wAIHA.
* Presence of unacceptable side effect(s) or toxicity associated with rilzabrutinib such that there is an unfavorable risk-benefit assessment for continued treatment with rilzabrutinib in the opinion of the Investigator and/or Sponsor.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Part A: Proportion of participants with overall hemoglobin response | By Week 24 in Part A
  Response is defined as an increase in hemoglobin (Hb) by ≥2 g/dL from baseline and an absence of transfusion in the last 7 days, without biochemical resolution of hemolysis at the time response is achieved and an absence of rescue medications during the last 4 weeks.
  Complete Response is defined as hemoglobin ≥11 g/dL (women) or ≥12 g/dL (men), no evidence of hemolysis (normal bilirubin, lactate dehydrogenase (LDH) , haptoglobin, and reticulocytes), and absence of transfusion in the last 7 days and an absence of rescue medications during the last 4 weeks.
Part B: Proportion of participants who maintain durable response achieved during Part A or achieve a durable response during Part B and have a hemoglobin response | By Week 50 in Part B
  Durable response (Part B) is defined as Hb level ≥10 g/dL with an increase from baseline (Part A) of ≥2 g/dL on three consecutive scheduled visits during Week 24 to Week 50; with absence of transfusion and no rescue medication during the period of 3 consecutive visits and for at least 7 days (transfusions) and 4 weeks (rescue medication) prior to the first consecutive visit.

SECONDARY OUTCOMES:
Proportion of participants with durable hemoglobin response | By Week 24 in Part A
  Durable response (Part A) is defined as Hb level ≥10 g/dL with an increase from baseline of ≥2 g/dL on three consecutive evaluable visits during the 24-week treatment period; with absence of transfusion and no rescue medication during the period of 3 consecutive visits and for at least 7 days (transfusions) and 4 weeks (rescue medication) prior to the first consecutive visit.
Median time from baseline to first hemoglobin response | From Day 1 to Week 24 in Part A
Frequency of rescue therapy (any wAIHA-directed therapy other than predniso[lo]ne or transfusion) received | After Week 1 of treatment to Week 24 in Part A and Week 305 in Part B
Change from baseline in FACIT-Fatigue scale score | Until Week 24 in Part A and Week 305 in Part B
  The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) scale is a 13-item questionnaire used to assesses self-reported fatigue and its impact on daily activities and function.
Incidence of treatment emergent adverse events (TEAEs), serious TEAEs, adverse events of special interest (AESIs) | Until Week 24 in Part A and Week 305 in Part B
  Safety assessment including clinical laboratory evaluations, vital sign measurements and ECG

CONTACTS AND LOCATIONS:
Locations (27):
- United States (11):
  - The Oncology Institute of Hope & Innovation Site Number : 8400006, Cerritos, California
  - TOI Clinical Research LLC_ Cerritos_Investigational Site Number: 8400006, Cerritos, California
  - TOI Clinical Research LLC_Glendale_Investigational Site Number: 8400006, Glendale, California
  - TOI Clinical Research LLC_Long Beach_Investigational Site Number: 8400006, Long Beach, California
  - University of Southern California_Investigational Site Number: 8400009, Los Angeles, California
  - TOI Clinical Research LLC_Santa Ana_Investigational Site Number: 8400006, Santa Ana, California
  - The Lundquist Institute_Investigational Site Number: 8400005, Torrance, California
  - TOI Clinical Research LLC_ Whittier_Investigational Site Number: 8400006, Whittier, California
  - Georgetown University Hospital_Investigational Site Number: 8400003, Washington D.C., District of Columbia
  - Oncology & Hematology Associates of West Broward_Investigational Site Number: 8400002, Tamarac, Florida
  - Massachusetts General Hospital_Investigational Site Number: 8400001, Boston, Massachusetts
- Hanush-Krankenhaus_Investigational Site Number: 0400001, Vienna, Austria
- China (2):
  - Peking Union Medical College Hospital_Investigational Site Number: 1560002, Beijing
  - Institute of hematology&blood diseases hospital_Investigational Site Number: 1560003, Tianjin
- Odense Universitetshospital Hæmatologisk Forskningsenhed_Investigational Site Number: 2080001, Odense, Denmark
- Klinik für Hämatologie und Stammzellentransplantation_Investigational Site Number: 2760001, Essen, Germany
- Fejer Varmegyei Szent Gyorgy Egyetemi Oktato Korhaz_Investigational Site Number: 3480001, Székesfehérvár, Hungary
- Italy (3):
  - Ospedale Giuseppe Moscati_Investigational Site Number: 3800002, Avellino
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori"_Investigational Site Number: 3800003, Meldola
  - Ospedale Maggiore Policlinico_Investigational Site Number: 3800001, Milan
- Spain (4):
  - Hospital Universitario de Cruces_Investigational Site Number: 7240004, Barakaldo
  - Hospital Clinic de Barcelona_Investigational Site Number: 7240001, Barcelona
  - Hospital Universitario La Paz_Investigational Site Number: 7240003, Madrid
  - Hospital Universitario Virgen del Rocío_Investigational Site Number: 7240002, Seville
- United Kingdom (3):
  - Leeds Teaching Hospitals NHS Trust_Investigational Site Number: 8260001, Leeds
  - Barts Health NHS Trust_Investigational Site Number: 8260005, London
  - Imperial College Healthcare NHS Trust_Investigational Site Number: 8260002, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org